CLINICAL TRIAL: NCT05416138
Title: The Effects of Closed-loop TMS-EEG on Immediate Prefrontal Activity and Approach/Avoidance Behavior
Brief Title: Theta Phase-specific TMS to Modulate Prefrontal Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00016214
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Approach/Avoidance Behavior
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TMS over the left prefrontal cortex (Experimental): Transcranial magnetic stimulation (TMS) will be administrated with a figure-8 coil over the left dorsolateral prefrontal cortex (DLPFC) at the intensity of up to 120% of the individualized resting motor threshold (rMT). Stimulation will be performed during and for the duration of the cognitive test. Up to three TMS pulses will be delivered at the beginning of every test trial (each trial duration is 2-6 seconds). The total duration of the cognitive testing and stimulation per session is approximately 40 minutes (in 4 blocks with breaks in-between).
  Interventions: Device: Transcranial magnetic stimulation (TMS)
- TMS over the head vertex (Sham Comparator): Transcranial magnetic stimulation (TMS) will be administrated with a figure-8 coil over the head vertex at the intensity of up to 120% of the individualized resting motor threshold (rMT). Stimulation will be performed during and for the duration of the cognitive test. Up to three TMS pulses will be delivered at the beginning of every test trial (each trial duration is 2-6 seconds). The total duration of the cognitive testing per session is approximately 40 minutes (in 4 blocks with breaks in-between).
  Interventions: Device: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS) — TMS will be performed at either peaks or troughs of ongoing prefrontal theta oscillations (3-7 Hz) concurrently with the cognitive test at the beginning of every test trial. Theta oscillations will be monitored in real-time at the left dorsolateral prefrontal cortex using electroencephalography (EEG).

SUMMARY:
The purpose of this study is to evaluate the causal link between the phase of ongoing theta oscillations in the prefrontal cortex and approach/avoidance (Ap/Av) behavior in adults using theta phase-specific transcranial magnetic stimulation (TMS).

DETAILED DESCRIPTION:
Approach/avoidance (Ap/Av) behavior is a reliable marker of the emotional processes in the human brain and a robust predictor of mood disorders. Although existing scientific studies found a correlation between the approach/avoidance behavior and ongoing theta activity (3-7 Hz) in the left dorsolateral prefrontal cortex, the causal evidence of the phase-dependent role and strength of association between the prefrontal theta oscillations and approach/avoidance behavior are still unclear. Here, we will monitor brain oscillations in real-time non-invasively using electroencephalography during the approach/avoidance test and modulate theta peaks or troughs with transcranial magnetic stimulation. These data will provide novel understanding of the mechanisms of emotional processing in human brain.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years old.
2. Confident level of English language.

Exclusion Criteria:

1. Chronic condition that requires pharmacological treatment over the course of study participation.
2. Metallic or electric implant in the head, neck, or chest area or otherwise MRI-noncompatible implants.
3. History or evidence of seizures, head injuries with loss of consciousness, chronic neurological or mental disorder.
4. Pregnancy or breast-feeding.
5. History or evidence of alcohol or drug addiction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Opitz, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Full or partial access to the preprocessed data will be provided upon the request to the faculty / research staff of recognized research, medical, and educational institutions for educational and scientific purposes. The request should be sent via an institutional email and will be stored with the study materials. The request should include a short description of the scientific or educational aims.
Time Frame: Data will be shared only upon request after the study has ended (within 6 months).
Access Criteria: To receive access, the study investigators need to be contacted via an institutional e-mail including a short description of the scientific or educational aims.

RESULTS

PARTICIPANT FLOW:
Groups:
- TMS Over the Prefrontal Cortex Followed by TMS Over the Head Vertex.: Transcranial magnetic stimulation (TMS) was first applied to the left dorsolateral prefrontal cortex (Condition 1) and then to the vertex of the head (Condition 2) at an intensity of up to 120% of the individualized resting motor threshold. During both conditions, participants performed the Approach/Avoidance task, which included the presentation of emotional stimuli. Each stimulus was accompanied by a simultaneous burst of TMS pulses, synchronized to either the peaks or troughs of the participant's left prefrontal theta waves (in randomized, interleaved order). Participants responded to each stimulus with a joystick movement (which should have been either congruent or incongruent as per the task hint, in randomized, interleaved order). The primary outcome measure was the difference in responses during TMS synchronized to theta wave peaks versus troughs.
- TMS Over the Head Vertex Followed by TMS Over the Prefrontal Cortex.: Transcranial magnetic stimulation (TMS) was first applied to the vertex of the head (Condition2) and then to the left dorsolateral prefrontal cortex (Condition 1) at an intensity of up to 120% of the individualized resting motor threshold. During both conditions, participants performed the Approach/Avoidance task, which included the presentation of emotional stimuli. Each stimulus was accompanied by a simultaneous burst of TMS pulses, synchronized to either the peaks or troughs of the participant's left prefrontal theta waves (in randomized, interleaved order). Participants responded to each stimulus with a joystick movement (which should have been either congruent or incongruent as per the task hint, in randomized, interleaved order). The primary outcome measure was the difference in responses during TMS synchronized to theta wave peaks versus troughs.
Period: Overall Study
Arm/Group | TMS Over the Prefrontal Cortex Followed by TMS Over the Head Vertex. | TMS Over the Head Vertex Followed by TMS Over the Prefrontal Cortex.
Started | 13 | 13
Completed | 11 | 12
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All 26 participants consented in this study
Arm/Group | All Participants
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Reaction Times in the Approach/Avoidance Test
Description: Reaction time (in milliseconds) in the Approach/Avoidance task during transcranial magnetic stimulation (TMS). TMS was synchronized to either the peaks or troughs of the participant's left prefrontal theta waves, in a randomized and counterbalanced order. The preregistered primary outcome measure is the average difference in reaction times between peak- and trough-synchronized stimulation stimuli. This statistical contrast specifically highlights the role of theta phase in phase-aligned stimulation.
Time Frame: During the stimulation/task for each condition (approximately 6 minutes per run, 4 runs per condition).
Population: Cross-over study - all participants were in both arms at different timepoints
Measure: Median (Standard Error); unit: milliseconds
Groups:
- TMS Over the Left Prefrontal Cortex: Transcranial magnetic stimulation (TMS) will be administrated with a figure-8 coil over the left dorsolateral prefrontal cortex (DLPFC) at the intensity of up to 120% of the individualized resting motor threshold (rMT).
  Stimulation will be performed during and for the duration of the cognitive test. Up to three TMS pulses will be delivered at the beginning of every test trial (each trial duration is 2-6 seconds). The total duration of the cognitive testing and stimulation per session is approximately 40 minutes (in 4 blocks with breaks in-between).
  Transcranial magnetic stimulation (TMS): TMS will be performed at either peaks or troughs of ongoing prefrontal theta oscillations (3-7 Hz) concurrently with the cognitive test at the beginning of every test trial. Theta oscillations will be monitored in real-time at the left dorsolateral prefrontal cortex using electroencephalography (EEG).
- TMS Over the Head Vertex: Transcranial magnetic stimulation (TMS) will be administrated with a figure-8 coil over the head vertex at the intensity of up to 120% of the individualized resting motor threshold (rMT). Stimulation will be performed during and for the duration of the cognitive test. Up to three TMS pulses will be delivered at the beginning of every test trial (each trial duration is 2-6 seconds). The total duration of the cognitive testing per session is approximately 40 minutes (in 4 blocks with breaks in-between). Transcranial magnetic stimulation (TMS): TMS will be performed at either peaks or troughs of ongoing prefrontal theta oscillations (3-7 Hz) concurrently with the cognitive test at the beginning of every test trial. Theta oscillations will be monitored in real-time at the left dorsolateral prefrontal cortex using electroencephalography (EEG).
Arm/Group | TMS Over the Left Prefrontal Cortex | TMS Over the Head Vertex
Number analyzed (Participants) | 23 | 23
milliseconds | 36.8 (16.3) | 12.4 (21.2)

2. Secondary Outcome: Amplitude of TMS Evoked Potentials
Description: Amplitude of transcranial magnetic stimulation (TMS)-evoked potentials (in microvolts) in ongoing electroencephalography (EEG) in the left prefrontal cortex during the TMS synchronized to either peaks or troughs of the participant's left prefrontal theta waves. The preregistered secondary outcome measure is the average difference in early absolute evoked potentials between peak- and trough-synchronized stimulation epochs. This statistical contrast specifically highlights the phase-specific effect of theta phase-aligned stimulation.
Time Frame: During the stimulation/task for each condition (approximately 6 minutes per run, 4 runs per condition).
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | TMS Over the Left Prefrontal Cortex | TMS Over the Head Vertex
Number analyzed (Participants) | 23 | 23
microvolts | 1.3 (1.9) | 0.2 (1.1)

ADVERSE EVENTS:
Time Frame: During the visit that included TMS procedures (4 hours)
Groups:
- TMS Over the Prefrontal Cortex Followed by TMS Over the Head Vertex.: Transcranial magnetic stimulation was first applied to the left dorsolateral prefrontal cortex (condition 1) and then to the head vertex (condition 2) at an intensity of up to 120% of the individualized resting motor threshold. During both conditions, the brain state during the stimulation (peaks vs. troughs of the participant's prefrontal theta wave) and the task stimuli (congruent vs. incongruent) were randomized and counterbalanced.
- TMS Over the Head Vertex Followed by TMS Over the Prefrontal Cortex.: Transcranial magnetic stimulation was first applied to the head vertex (condition 2) and then to the left dorsolateral prefrontal cortex (condition 1) at an intensity of up to 120% of the individualized resting motor threshold. During both conditions, the brain state during the stimulation (peaks vs. troughs of the participant's prefrontal theta wave) and the task stimuli (congruent vs. incongruent) were randomized and counterbalanced.
Arm/Group | TMS Over the Prefrontal Cortex Followed by TMS Over the Head Vertex. | TMS Over the Head Vertex Followed by TMS Over the Prefrontal Cortex.
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT05416138/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT05416138/ICF_000.pdf